CLINICAL TRIAL: NCT01395498
Title: Prevalence of Positive DNA of Pneumocystis Jirovecii and of Cytomegalovirus in Bronchial Wash Fluid of Patients Undergoing Fiberoptic Bronchoscopy
Brief Title: Prevalence of Pneumocystis Jirovecii and of Cytomegalovirus in Bronchial Wash Fluid of Patients Undergoing Bronchoscopy
Acronym: PCP-CMV
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Michal Steinberg, Dr. Michal Shteinberg, Carmel Medical Center
Other Study IDs: CMC-11-0009-CTIL
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Patients Scheduled for Bronchoscopy
Keywords: CMV; PCP; bronchoalveolar lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples of bronchoalveolar lavage fluid and blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fiberoptic bronchoscopy: patients undergoing fiberoptic bronchoscopy who are not immunocompromized and in whom an opportunistic infection is not suspected.
  Interventions: Other: laboratory testing of PCP and CMV genetic material

INTERVENTIONS:
Other: laboratory testing of PCP and CMV genetic material — laboratory testing of PCP and CMV DNA in bronchoalveolar lavage fluid, CMV PCR in blood+ serology in patients with positive BAL.

SUMMARY:
The purpose of this study is to determine the incidence of the "carriage" state (asymptomatic colonization) with Pneumocystis Jirovecii (Pneumocystic Carinii Pneumonia, PCP) and Cytomegalovirus (CMV)in the human lung. These are pathogens causing pneumonia in patients with suppressed immune system, but not known to cause disease in otherwise normal people. The investigators hypothesis is that a carriage state exists for these two pathogens. To test this hypothesis the investigators will examine bronchoalveolar lavage fluid for genetic material of these two pathogens. The study population will be patients undergoing fiberoptic bronchoscopy and lavage for indications other than diagnosis of a presumed opportunistic infection.

DETAILED DESCRIPTION:
Both Pneumocystis Jirovecii (Pneumocystic Carinii Pneumonia, PCP) and Cytomegalovirus (CMV) are opportunistic pathogens known to cause infection in patients with impaired immune systems. PCP is a frequent pathogen causing respiratory tract infections in Acquired Immune Deficiency (AIDS) patients, but may also cause infection in other immunecompromised hosts. CMV is a causative agent of pneumonia mostly in transplant recipients.

For CMV pneumonia to be diagnosed in a patient with clinical signs of pneumonia, it is necessary to demonstrate the presence of the virus by its isolation, histopathologic testing, immunohistochemical analysis, or in situ hybridization. Detection of viral DNA in respiratory secretions (eg. Bronchial wash) may be too sensitive and is considered insufficient for diagnosis. However, the diagnostic methods are either not commonly performed or, in the case of histopathology, may risk severely ill patients. It is not known how often viral DNA is indeed detected in respiratory secretions of immunocompetent and immunocompromized hosts.

As for PCP, it is not known whether an asymptomatic carriage state exists for this pathogen. It has been suggested that PCP may be found in bronchial washings of asymptomatic patients, mostly corticosteroid- treated , and pregnant women. This finding has not been confirmed by other investigators, nor is it known what the prevalence of PCP colonization is in Israel. If PCP colonization is common, detection of PCP DNA in bronchial wash may represent colonization, not infection, and may mask true infection by an unidentified pathogen. Thus, it is of importance to define the prevalence of PCP in respiratory secretions in our population.

Bronchial washing is a procedure routinely performed during Fiberoptic Bronchoscopy, which includes the instillation of 10-20 ml sterile saline solution into a segmental or subsegmental bronchus. It is a safe procedure, which may rarely result in fever up to 38.5 up to a few hours after the procedure. Patients hypoxemic at room air (O2 Sat <90%) will be excluded from this study.

Study Procedures:

In order to assess the prevalence of detection of PCP and CMV DNA in respiratory secretions, we propose to prospectively perform polymerase chain reaction (PCR) analysis of PCP and of CMV DNA in bronchial wash obtained during bronchoscopy. In order to correlate CMV findings to blood antigenemia and viremia, 5 ml of blood will be drawn for analysis of CMV antibodies (IgG) and CMV DNA (PCR analysis). Blood will be drawn during insertion of venous access routinely performed for sedation during the procedure.

Patients will be those undergoing scheduled Fiberoptic Bronchoscopy for other indications and not as part of the study protocol. Indication for Fiberoptic Bronchoscopy will be recorded, as well as any associated medical condition and chronic medication

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Fiberoptic Bronchoscopy for any indication and signing an informed consent form.

Exclusion Criteria:

* Hypoxemia < 90% at Room air

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients cared for in the pulmonology outpatients clinic and for whom a fiberoptic bronchoscopy is indicated.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Adir, MD, Study Director — Pulmonology Institute, Carmel Medical Center
Locations (1):
- Pulmonology Institute, Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shteinberg M, Shaked-Mishan P, Kinarti A, Abramovitch A, Amital A, Jacobi A, Kolup Feldmann AE, Shiner M, Gershtein V, Weber G, Adir Y. Asymptomatic carriage of Pneumocystis jirovecii and cytomegalovirus in lungs of immunocompetent patients. Lung. 2014 Dec;192(6):875-9. doi: 10.1007/s00408-014-9644-z. Epub 2014 Sep 9. PMID 25201088